CLINICAL TRIAL: NCT02006147
Title: Phase I/II Trial of TLC399 (ProDex) in Patients With Macular Edema Due to Retinal Vein Occlusion (RVO)
Brief Title: Phase 1 Open-label Study to Evaluate Efficacy and Tolerability of TLC399 in Patients With Macular Edema Due to RVO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TLC399.1
Record Dates: First submitted 2013-11-13; First posted 2013-12-10 (Estimated); Results first posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Central Retinal Vein Occlusion With Macular Edema; Branch Retinal Vein Occlusion With Macular Edema
Keywords: Macular Edema; RVO
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TLC399 (Group 1) (Experimental): TLC399 is manufactured with the proprietary lipid formulation in lyophilized form (BioSeizer) for the reconstitution with the aqueous DSP.
  Interventions: Drug: TLC399
- TLC399 (Group R1) (Experimental): TLC399 is manufactured with the proprietary lipid formulation in lyophilized form (BioSeizer) for the reconstitution with the aqueous DSP.
  Interventions: Drug: TLC399
- TLC399 (Group 2) (Experimental): TLC399 is manufactured with the proprietary lipid formulation in lyophilized form (BioSeizer) for the reconstitution with the aqueous DSP.
  Interventions: Drug: TLC399
- TLC399 (Group 3) (Experimental): TLC399 is manufactured with the proprietary lipid formulation in lyophilized form (BioSeizer) for the reconstitution with the aqueous DSP.
  Interventions: Drug: TLC399

INTERVENTIONS:
Drug: TLC399 — Dose-escalation Study from 100 mM PL (20 µL) with 0.24 mg DSP to 100 mM PL (20 µL) with0.36 mg DSP to 100 mM PL (20 µL) with 0.6 mg DSP to 50 mM PL (10 µL) with 0.6 mg DSP.
  Other Names: TLC399 (BioSeizer)

SUMMARY:
To determine whether TLC399 (ProDex) provides an ideal, safe, long-acting, dexamethasone sodium phosphate (DSP) delivery system for the treatment of macular edema due to retinal vein occlusion (RVO).

DETAILED DESCRIPTION:
<Part 1> An open-label, sequential dose escalation part to determine the DLT of TLC399 (ProDex) in patients with macular edema due to central retinal vein occlusion (CRVO) or branch retinal vein occlusion (BRVO). The safety results should be evaluated by Safety Monitor Committee regularly every 6 months and after last patient of each cohort completes DLT observation period. The SMC would advise or give permission for further dose escalation, de-escalation, or any study design adjustment. After the study drug administration, these patients will continue to be evaluated for efficacy and safety outcomes up to a period of 12 months unless the patient is withdrawn or discontinues the study.

* Group R1: 0.24 mg DSP with 100 mM PL (20 µL)
* Group 1: 0.36 mg DSP with 100 mM PL (30 µL)
* Group 2: 0.6 mg DSP with 100 mM PL (50 µL)
* Group 3: 0.6 mg DSP with 50 mM PL (50 µL)

<Part 2> An open-label, single-arm design to investigate the use of TLC399 (ProDex) in patients with macular edema due to CRVO or BRVO in one dose level selected from Part 1. The enrollment of subjects for analysis will include approximately 20 patients in total, inclusive of Part 1 and Part 2 for the selected dose group. The safety and efficacy outcomes will be assessed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, > 20 years of age.
* Patients with macular edema due to CRVO or BRVO diagnosed within 36 months.
* BCVA score of 20/40 to 20/400 by chart ETDRS in the study eye.
* Mean central subfield thickness ≥350uM on Spectral/Fourier domain by OCT measurements in the study eye.
* Willing and able to comply with the study procedure and sign a written informed consent.

Exclusion Criteria:

* Macular edema due to diabetic retinopathy or other etiologies.
* Brisk afferent pupillary defect.
* Stroke or myocardial infarction within 3 months.
* Uncontrolled systemic disease, or poorly controlled hypertension, or poorly controlled diabetes.
* Any ocular condition that in the opinion of the Investigator would prevent a 15-letter gain in visual acuity.
* Presence of an epiretinal membrane in the study eye which is the primary cause of macular edema, or is severe enough to prevent gain in visual acuity despite reduction in macular edema.
* History of clinically significant IOP elevation in response to steroid treatment.
* History of glaucoma or optic nerve head change consistent with glaucoma damage, and/or glaucomatous visual field loss in both eyes.
* Active ocular hypertension ≥21mmHg or history of treated ocular hypertension in the study eye.
* Aphakia or presence of anterior chamber intraocular lens in the study eye.
* Active retinal neovascularization in the study eye.
* Active or history of choroidal neovascularization in the study eye.
* History of central serous chorioretinopathy in either eye.
* Presence of rubeosis iridis in the study eye.
* Any active ocular infection in either eye.
* History of herpetic ocular infection in the study eye or adnexa.
* Presence of active or inactive toxoplasmosis in either eye.
* Presence of visible scleral thinning or ectasia in the study eye.
* Media opacity in the study eye that precludes clinical and photographic evaluation.
* Intraocular surgery in the stydy eye within 6 months.
* History of pars plana vitrectomy, radial optic neurotomy, or sheathotomy in the study eye.
* Anticipated need for ocular surgery in the study eye during the 12-months study period.
* Use of hemodilution for the treatment of RVO within 3 months.
* Use of any intraocular anti-VEGF therapy in the study eye.
* Use of laser of any type in the study eye within 3 months.
* Previous use of intravitreal steroids in the study eye within 6 months.
* Periocular depot of steroids to the study eye within 1 month.
* Use of systemic sterois, or warfarin/heparin within 1 month.
* Use of immunosuppressants, immunomodulators, antimetabolites, and/or alkylating agents within 6 months.
* BCVA score <34 letters in the non-study eye.
* Known allergy or hypersensitivity to the study medication or its components.
* Known allergy or contraindication to the use of fluorescein or povidone iodine or contraindication to pupil dilation in either eye.
* Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception.
* Current enrollment in an investigational drug or device study or participation in such a study within 90 days.
* Patient has a condition or is in a situation which will interfere with the patient's ability to comply with the dosig and visit schedules and the protocol evaluations or may not suitable for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (6):
- Taiwan (6):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Chang-hua
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Groups:
- TLC399 (Group 1): 0.36 mg Dexamethasone Sodium Phosphate with 100 mM Phospholipid
- TLC399 (Group R1): 0.24 mg Dexamethasone Sodium Phosphate with 100 mM Phospholipid
- TLC399 (Group 2): 0.6 mg Dexamethasone Sodium Phosphate with 100 mM Phospholipid
- TLC399 (Group 3): 0.6 mg Dexamethasone Sodium Phosphate with 50 mM Phospholipid
Period: Overall Study
Arm/Group | TLC399 (Group 1) | TLC399 (Group R1) | TLC399 (Group 2) | TLC399 (Group 3)
Started | 5 | 9 | 0 | 0
Completed | 3 | 7 | 0 | 0
Not Completed | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Withdrawal by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population was based on the Safety Populaiont who exposed to study treatment, either complete or partial.
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC399 (Group 1) | TLC399 (Group R1) | TLC399 (Group 2) | TLC399 (Group 3) | Total
Number analyzed (Participants) | 4 | 9 | 0 | 0 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.4) | 65.8 (16.2) |  |  | 64.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 |  |  | 8
  Male | 0 | 5 |  |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 4 | 9 |  |  | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 0 | 0 |  |  | 0
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 4 | 9 |  |  | 13
Macular edema by retinal vein occlusion [Count of Participants; unit: Participants]
  Branch retinal vein occlusion | 3 | 7 |  |  | 10
  Central retinal vein occlusion | 1 | 2 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Dose-limiting Toxicity (DLT)
Description: Ocular AEs
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TLC399 (Group 1) | TLC399 (Group R1)
Number analyzed (Participants) | 4 | 9
Participants | 1 | 0

2. Primary Outcome: Part 2: Safety Assessment: Number of SAEs and Treatment-related Severe AEs
Description: Number of SAEs and treatment-related severe AEs
Time Frame: Up to 1 year
Measure: Number; unit: Number of events
Arm/Group | TLC399 (Group 1) | TLC399 (Group R1)
Number analyzed (Participants) | 4 | 9
Number of events
  Number of SAE | 2 | 5
  Number of Treatment-related severe AE | 0 | 5

ADVERSE EVENTS:
Time Frame: 14 days (screeing) + 1 year
Arm/Group | TLC399 (Group 1) | TLC399 (Group R1)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/9
Other Adverse Events (participants affected / at risk) | 4/4 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TLC399 (Group 1) (N=4) | TLC399 (Group R1) (N=9)
Head Injury With Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ocular Hypertension (Eye disorders) | 1 | 0
Intraocular Pressure Increased (Investigations) | 0 | 1
Prolong Vitreous Opacity (Eye disorders) | 0 | 1
IOP Elevation (Investigations) | 0 | 1
More than 30 Letters Visual Acuity Reduction from Baseline of BCVA (Eye disorders) | 0 | 1
Increased Intraocular Pressure (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TLC399 (Group 1) (N=4) | TLC399 (Group R1) (N=9)
Vitreous opacities (Eye disorders) | 4 | 6
Visual acuity reduced (Eye disorders) | 2 | 5
Conjunctival haemorrhage (Eye disorders) | 2 | 2
Corneal oedema (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 2
Macular oedea (Eye disorders) | 0 | 2
Ocular hypertension (Eye disorders) | 2 | 0
Retinal thickening (Eye disorders) | 1 | 1
Abnormal sensation in eye (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 1 | 0
Conjunctival follicles (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye opacity (Eye disorders) | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 1 | 0
Hyalosis asteroid (Eye disorders) | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 1
Retinal disorder (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Vitreous haze (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Sensation of foreign body (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 5
Alanine aminotransferase increase (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Intraocular pressure decreased (Investigations) | 0 | 1
Optic nerve cup/disc ratio increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Visual field defect (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT02006147/Prot_SAP_000.pdf